CLINICAL TRIAL: NCT02723942
Title: Chimeric Antigen Receptor-Modified T Cell (CAR-T) Immunotherapy for Hepatocellular Carcinoma (HCC) Targeting Glypican-3 (GPC3)
Brief Title: CAR-T Cell Immunotherapy for HCC Targeting GPC3
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Project terminated due to revision of local regulations
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T for GPC3+ HCC
Record Dates: First submitted 2016-03-20; First posted 2016-03-31 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: GPC3 Positive Hepatocellular Carcinoma; CAR-T Cell Immunotherapy
Keywords: glypican-3(GPC3); chimeric antigen receptor-modified T cell(CAR-T); hepatocellular carcinoma(HCC)
MeSH Terms: conditions — Simpson-Golabi-Behmel syndrome; Carcinoma, Hepatocellular | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAR-T cell immunotherapy (Experimental): Enrolled patients will receive CAR-T cell immunotherapy with a novel specific Chimeric antigen receptor aiming at GPC3 antigen by infusion.
  Interventions: Biological: CAR-T cell immunotherapy
- no intervention (No Intervention): no intervention

INTERVENTIONS:
Biological: CAR-T cell immunotherapy — This CAR-T cell immunotherapy with a novel specific Chimeric antigen receptor aiming at GPC3 antigen.
  Arms: CAR-T cell immunotherapy

SUMMARY:
The purpose of this study is to preliminarily evaluate the safety and efficacy of CAR-T cell immunotherapy for GPC3 positive hepatocellular carcinoma.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) is a recombinant receptor with both antigen-binding and T cell activating functions. Chimeric antigen receptor T cell Immunotherapy has more advantages compared with conventional immunotherapy, especially in dealing with patients of hematologic malignancies and solid malignant tumors.This study design a novel specific Chimeric antigen receptor targeting glypican-3(GPC3) antigen.After CAR-T cell infusion,At periodic intervals, the investigators will evaluate clinical symptoms Improved conditions of this disease.Through this study,the investigators will evaluate the safety and efficacy of CAR-T cell immunotherapy in treating with GPC3 positive malignant glioma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-70 years.
2. Gender:both.
3. GPC3 high expression hepatocellular carcinoma patients.
4. Non diffuse hepatocellular carcinoma，no extrahepatic metastasis or portal vein vascular invasion.
5. Degree of liver cirrhosis：class A or class B 7 according to Child-puge grading standard.
6. Routine blood test：white blood cell count（WBC)>=3×10^9/L, Lymphocyte percentage>=15%, hemoglobinHbo（Hb）>=90g/L, prothrombin time（PT） prolongation<=50% normal value, Cluster of differentiation 3(CD3) positive T cell count>=0.8×10^9/L.
7. Liver and Pancreatic function：Alanine aminotransferase/Aspartate transaminase(ALT/AST)<=5 times of the normal value, total bilirubin(TBiL)<=3.0mg/dL, albumin(ALB)>=35g/L, prothrombin time(PT):International Normalized Ratio(INR)<=1.7 or prothrombin time(PT) prolongation<=4s, Serum lipase<=1.5 times of the normal value, Serum amylase<=1.5 times of the normal value.
8. Renal function：Serum creatinine(SCr)<=221μmol/L(2.5mg/L).
9. Karnofsky Performance Status(KPS)>=60；Expected survival time>=12 weeks.
10. Peripheral venous access ；no contraindication of lymphocyte separation.
11. No other serious complications.
12. Voluntarily signed informed consent.

Exclusion Criteria:

1. Pregnant and lactating women.
2. Lymphocyte separation or peripheral venous access cannot be performed in patients .
3. Patients in the active stage of infection or with coagulation disorders.
4. Patients with a previous history of hepatic coma.
5. Patients with severe gastrointestinal ulcers or gastrointestinal bleeding.
6. Patients with organ transplantation or waiting for organ transplantation.
7. Patients with anticoagulant therapy.
8. Patients with antiplatelet therapy.
9. Serum sodium(Na)<125 mmol/L.
10. Serum potassium(K)<3.5 mmol/L(except patients up to the standards after the use of supplements).
11. Patients with organ failure：

    1. cardiac function：level three or above according to New York Heart Association (NYHA) criteria.
    2. liver function:class C or above according to Child-puge grading standard.
    3. renal function:Chronic kidney disease(CKD) phase 4 or more; renal insufficiency phase Ⅲ or more.
    4. pulmonary function：severe respiratory failure symptoms, involving other organs.
    5. Brain function:central nervous system abnormalities or disturbance of consciousness.
12. Patients with non controlled infectious diseases,for example,HIV positive, syphilis, hepatitis A, hepatitis B, hepatitis C, hepatitis E virus (HEV) positive etc.
13. Patients used corticosteroids or other immunosuppressive agents in the past 4 weeks.
14. Patients with autoimmune disease.
15. Patients with previous history of gene therapy.
16. The actual transfection rate of T cells was lower than 30% or the proliferation was less than 5 times after costimulation.
17. Patients participated in other drug trials in the past 4 weeks.
18. Patients received radiation treatment in the past 4 weeks.
19. Patients do not meet the criteria above.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Radiological assessment | 3 months
  Radiological assessment of the therapeutic effect by systemic or local computed Tomography(CT) or positron emission tomography scan.

SECONDARY OUTCOMES:
The safety of CAR-T cell immunotherapy (adverse events) | 4 weeks
  After CAR-T cell infusion,we will observe the potential adverse events related to the T-cell infusion such as high fever,jaundice, kidney failure and so on.
Peripheral blood tumor markers | 3 months
  tested regularly to reflect the role of the Chimeric Antigen Receptor-Modified T Cell in the removal of residual tumor cells.
CAR-T cell testing | 3 months
  The level of CAR-T cells will be tested regularly by Real-time Quantitative Polymerase Chain Reaction Detecting System(qPCR) or Flow cytometry to evaluate the proliferation in vivo and long-term survival.

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China